CLINICAL TRIAL: NCT03600337
Title: An Integrated Self-Management Intervention for Adolescents With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Fordham University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Cara Young, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-08-0024; 5P30NR015335 (NIH)
Record Dates: First submitted 2018-07-02; First posted 2018-07-26 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: PCOS

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Condition (Experimental): Working to Optimize Wellness in Teens with PCOS
  Interventions: Behavioral: Working to Optimize Wellness in Tees with PCOS (WOW)
- Control Condition (No Intervention): Participants in this arm will receive treatment as usual and will be given the intervention after 1 month assessments are completed for the intervention group

INTERVENTIONS:
Behavioral: Working to Optimize Wellness in Tees with PCOS (WOW) — 5 week, 75 minutes weekly, integrated mindfulness-based mental and physical health promotion intervention
  Arms: Experimental Condition

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common female endocrine disorder, affecting 7%-18% of reproductive-age women. Women with PCOS are at increased risk for a number of adverse physical and mental health outcomes. Often diagnosed during the challenging developmental period of adolescence (ages 14-18), current clinical practice guidelines fail to consider the life-long nature of effective PCOS self-management through sustained healthy lifestyle habits and may, in fact, contribute to maladaptive patterns of unsustainable strategies for weight loss in adolescents. The investigators are testing an integrated mindfulness-based healthy lifestyle intervention for adolescents with PCOS (Working to Optimize Wellness in Teens with PCOS [WOW]). The purpose of this study is to obtain data supporting preliminary efficacy of WOW on biological and mental health outcomes with adolescents diagnosed with PCOS.

DETAILED DESCRIPTION:
Innovative approaches to addressing the unique physical and mental health needs of adolescents with PCOS are needed. In response to this need, the investigators have developed an integrated mindfulness-based healthy lifestyle intervention for adolescents with PCOS (Working to Optimize Wellness in Teens with PCOS [WOW] through an iterative process of serial focus groups with adolescents and parents of adolescents with PCOS guided by the Individual and Family Self-Management Theory (IFSMT). In this pilot randomized control trial (RCT), 40 adolescents aged 14-18 years will be recruited to participate in the 5-week Working to Optimize Wellness in Teens with PCOS (WOW) intervention (N=20) or a waitlist-control condition (n=20). All participants will receive treatment as usual. Participants will meet weekly for 75-90 minutes for five weeks. Data collection will occur at 3 time points: Baseline data (T1) will be collected from all participants immediately following the informed consent process, Time 2 (T2) data will be collected immediately post-intervention, and Time 3 (T3) data will be collected one-month post-intervention. The waitlist- control condition will receive the intervention immediately following the one-month post-intervention data collection period. Following completion of the self-report measures at T3, individual exit interviews will be conducted with a subset of participants (N=10) from the WOW condition.

The primary aims of this research study are:

1. To conduct a pilot RCT with 40 adolescents (ages 14-18) diagnosed with PCOS comparing WOW (n=20) to a wait-list control condition (n=20), and conduct individual exit-interviews to further refine WOW. The investigators expect to determine:

a. Preliminary effects of WOW vs. wait-list control on blood pressure, fasting insulin, hemoglobin A1C, nutrition self-efficacy, physical activity, medication adherence, psychological well-being (i.e., depressive/anxiety symptoms, perceived stress, self-esteem) and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* adolescent age 14-23 years,
* diagnosis of PCOS, OR obesity AND secondary amenorrhea, OR excessive and frequent menstruation and
* ability to provide informed consent.

Exclusion Criteria:

* inability to commit to attending all intervention sessions
* unable to provide written informed consent/assent
* loss of a loved one within the last year, or
* history of post-traumatic stress disorder

Ages: 14 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Change in psychological distress | Immediately post-intervention
  The Depression, Anxiety, and Stress Scale is a 21-item standardized scale that assess symptoms of depression, anxiety, and perceived stress. Participants rate each item from 0=Did not apply to me at all to 3=Applied to me very much or most of the time. All items are summed for a possible range from 0-63 with higher scores indicating higher levels of psychological distress.
Change in health related quality of life | Immediately post-intervention
  The Child Health Questionnaire-Child Self-Report Form is an 87-item measure consisting of 12 summed subscales assessing unique physical and psychosocial domains. Items are scored from 0 to 100 with higher scores indicating better quality of life

SECONDARY OUTCOMES:
Change in Diet self-efficacy | Immediately post-intervention, 1-month post-intervention
  The Diet Self-Efficacy Scale is an 11-item standardized measure assessing self-efficacy for healthy nutrition choices in three domains, (a) high caloric food temptation, (b) social and internal factors, and (c) negative emotional events. For each item, participants select their level of confidence from 0=Not at all confident to 4= Very confident. Item scores are summed for a possible score range from 0 (very little diet self-efficacy) to 44 (very high diet self-efficacy).
Change in Physical activity self-efficacy | Immediately post-intervention, 1-month post-intervention
  The PACE Adolescent Physical Activity Survey is a 50-item standardized measure that assesses adolescents' stage of change, self-efficacy, family support, and peer support for physical activity. Self-efficacy is assessed with 7 items rated from 1=I'm sure I can't to 5=I'm sure I can. The mean of these 7 items will be used to assess physical activity self-efficacy immediately post-intervention and again at 1-month post-intervention with a possible score range from 1 to 7 and higher scores indicating higher self-efficacy for physical activity.
Change in self-esteem | Immediately post-intervention
  The Rosenberg Self-Esteem Scale is a 10-item scale that measures an individual's self-esteem. Participants rate each item from 3=Strongly Agree to 0=Strongly Disagree. Scores for the 10 items are summed for a possible score from 0 to 40 with higher scores indicating higher self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Cara C Young, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States